CLINICAL TRIAL: NCT02283372
Title: Prospective Phase I Study of Nab-Paclitaxel Plus Gemcitabine With Concurrent MR-Guided IMRT in Patients With Locally Advanced Pancreatic Cancer
Brief Title: Nab-Paclitaxel Plus Gemcitabine With Concurrent MR-Guided IMRT in Patients With Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201412038
Record Dates: First submitted 2014-10-24; First posted 2014-11-05 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- nab-Paclitaxel + Gemcitabine + IMRT (Experimental): * Prior to initiation of chemoradiation, patients will undergo 1 full cycle of gemcitabine and nab-paclitaxel on Days 1, 8, and 15 of a 28-day cycle.
  * Both gemcitabine and nab-paclitaxel will be given intravenously on an outpatient basis during the one-month lead-in period and during Weeks 1 and 2 (and, if enrolled to Dose Level or 2, Weeks 4 and 5) of radiotherapy. There may be up to 21 days between the last dose of lead-in chemotherapy (given on Day 15) and initiation of chemoradiation (inclusive of the week following Day 15, the fourth week of the lead-in cycle (an off-week), and an additional week following that).
  * Intensity modulated radiation (IMRT) - the prescribed dose will range from 40-67.5 Gy over 15 to 25 fractions.
  Interventions: Drug: nab-Paclitaxel; Drug: Gemcitabine; Radiation: Intensity modulated radiation

INTERVENTIONS:
Drug: nab-Paclitaxel
  Other Names: Abraxane; Albumin-bound paclitaxel
Drug: Gemcitabine
  Other Names: Gemzar®
Radiation: Intensity modulated radiation
  Other Names: IMRT

SUMMARY:
A phase I study to evaluate safety of gemcitabine with nab-paclitaxel and concurrent IMRT for locally advanced and borderline resectable pancreatic cancer. The goal of this study is to evaluate if a chemotherapy regimen that provides superior systemic efficacy may be safely delivered and enhance efficacy of tumor directed radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced adenocarcinoma of the pancreas that is considered unresectable or borderline resectable based on institutional standardized criteria of unresectability or medical inoperability. Patients with and without regional adenopathy are eligible.
* Prior systemic chemotherapy allowed. It is anticipated and suggested that most patients enrolled on study will have received a minimum of approximately 2 months of systemic therapy according to routine institutional practices. The patient must also be felt by the treating medical oncologist and radiation oncologist to be a candidate for treatment with gemcitabine/nab-paclitaxel chemoradiotherapy.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,000/mcl
  * Platelets ≥ 100,000/mcl
  * Hemoglobin ≥ 9.0 g/dL
  * Total bilirubin ≤ 1.5 x ULN
  * AST(SGOT)/ALT(SGPT) ≤ 1.5 x IULN
  * Serum creatinine ≤ 1.5 mg/dL or calculated CrCL>60mL/min using Cockcroft and Gault formula
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Distant metastatic disease, including known brain metastases.
* History of prior malignancy is acceptable, but prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields is not allowed.
* Currently receiving any other investigational agents.
* Major surgery within 4 weeks prior to first study drug administration.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine or nab-paclitaxel or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding. Patient must have a negative pregnancy test within 14 days of study entry.
* Known HIV-positivity on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with gemcitabine and nab-paclitaxel. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2019-04-18 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Completion of toxicity follow-up for all patients (up to 32 months)
  For the toxicity endpoint purposes of this trial, the patient will be followed from start of treatment until the patient completes 60 days of follow-up from the start of radiation therapy, has a dose-limiting toxicity (DLT), or is lost to follow-up.

SECONDARY OUTCOMES:
Rate of conversion of patients with locally advanced pancreatic cancer or borderline resectable to resectable | 1 year
Local control (Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) | 1 year
  Local control is absence of tumor progression.
  Response and progression will be evaluated in this study using the new international criteria proposed by the revised
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Progression-free survival (PFS) | 1 year
Overall survival (OS) | 1 year
Quality of life as measured by the EORTC QLQ-C30 | 3 months after completion of treatment (up to 18 weeks)
  The EORTC QLQ-C30 questionnaire will be utilized.
Frequency of RT adaptation based on MR guidance | 3 months after completion of treatment (up to 18 weeks)
  The rate at which a change or adaptation to the patient's plan is made based on significant change in anatomy observed on localization MRI. This is defined as [#of treatment adaptations required]/[total # of RT treatments]

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Kim, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu